CLINICAL TRIAL: NCT01407640
Title: Diagnosis and Physiopathology of Insulin Allergy (IA)
Brief Title: Diagnosis and Physiopathology of Insulin Allergy
Acronym: Allerdiab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P081223
Record Dates: First submitted 2011-06-28; First posted 2011-08-02 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Hypersensitivity; Immediate Hypersensitivity; Allergy
Keywords: Insulin allergy; adverse drug reaction; diabetes; type 1 hypersensitivity; immediate hypersensitivity; type 4 hypersensitivity; insulin analogs; intradermal testing; insulin antibody; mast cell; CD+ TCELL
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Hypersensitivity; Hypersensitivity, Immediate; Drug-Related Side Effects and Adverse Reactions; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Allergy tests
  Interventions: Procedure: Allergy tests

INTERVENTIONS:
Procedure: Allergy tests — 1/ to validate a diagnostic algorithm for patients presenting with possible allergy. 2/ to investigate immunogenetic profiles of patient with insulin allergy 3/ cellular mechanisms of IA

SUMMARY:
Insulin allergy (IA) is still observed even with recombinant human insulin and insulin analogs.

Obviously, the usual attitude facing an allergy, i. e. exclusion of the allergen, poses problems in face of IA because insulin is often vital for the patient. IA is thus a complex situation in which a rigorous diagnostic procedure to identify the exact allergen is necessary to propose a therapeutic answer; the purpose of the study is 1/ to validate a diagnostic algorithm for patients presenting with possible allergy. 2/ to investigate immunogenetic profiles of patient with insulin allergy 3/ cellular mechanisms of IA.

DETAILED DESCRIPTION:
Phenotype of the patient Investigation of allergy per intradermal testing using a wide range of insulin preparations Determination of immunologic and immunogenetic profile particularly CD4 + T cells and mast cells

ELIGIBILITY:
Inclusion criteria :

* Patients aged 18 years old and more with a written informed consent
* Experimental group : type 1 or type 2 diabetic patients with insulin allergy based on clinical criteria
* Active Comparator group: type 1 or type 2 diabetic patients insulin treated without insulin allergy

Exclusion criteria :

* Not willing participate
* Pregnancy
* Age below 18 years
* Severe Renal failure
* Severe Anaphylactic shock only for the experimental group
* No social security overture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

PRIMARY OUTCOMES:
Validation of cutaneous insulin tests | after 36 months
  Response of cutaneous insulin tests in patients with IA (Insulin Allergy) at study completion.

SECONDARY OUTCOMES:
Immunogenetic of patients with IA (Insulin Allergy) | after 36 months
  Immunogenetic of patients with IA (Insulin Allergy) at study completion Determination of insulin epitopes that are involved in IA at study completion Determination of isotypes of anti insulin antibodies and whether specific isotypes are associated with susceptibility / protection at study completion

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Sola-Gazagnes, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Background] Sola-Gazagnes A, Pecquet C, Berre S, Achenbach P, Pierson LA, Virmoux-Buisson I, M'Bemba J, Elgrably F, Moguelet P, Boitard C, Caillat-Zucman S, Laanani M, Coste J, Larger E, Mallone R. Insulin allergy: a diagnostic and therapeutic strategy based on a retrospective cohort and a case-control study. Diabetologia. 2022 Aug;65(8):1278-1290. doi: 10.1007/s00125-022-05710-9. Epub 2022 May 4. PMID 35505238
- [Background] Sola-Gazagnes A, Pecquet C, Radermecker R, Pietri L, Elgrably F, Slama G, Selam JL. Successful treatment of insulin allergy in a type 1 diabetic patient by means of constant subcutaneous pump infusion of insulin. Diabetes Care. 2003 Oct;26(10):2961-2. doi: 10.2337/diacare.26.10.2961. No abstract available. PMID 14514615
- [Background] Sola-Gazagnes A, Pecquet C. [Allergy to insulin in 2003]. Journ Annu Diabetol Hotel Dieu. 2004:161-79. No abstract available. French. PMID 15259314
- [Background] Sola-Gazagnes A, Pecquet C, M'Bemba J, Larger E, Slama G. Type I and type IV allergy to the insulin analogue detemir. Lancet. 2007 Feb 24;369(9562):637-8. doi: 10.1016/S0140-6736(07)60301-8. No abstract available. PMID 17321300